CLINICAL TRIAL: NCT02355769
Title: Multiparametric Assessment of Complex Pathophysiological Background of Heart Failure Deterioration - Relation to Treatment Effects and Prognosis
Brief Title: Complex Pathophysiological Background of Heart Failure Deterioration
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Paweł Krzesiński, Scientific Assistant, Military Institute od Medicine National Research Institute
Other Study IDs: WIM-0000000213
Record Dates: First submitted 2015-01-22; First posted 2015-02-04 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure
Keywords: heart failure; renal failure; prognosis; impedance cardiography
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Preventing heart failure (HF) deterioration is a great challenge for contemporary medicine. The progress course of HF is with increasing frequency of subsequent hospitalizations (approximately 30% of hospitalizations are the repeated ones). It is estimated that the costs of hospital stays constitute nearly 2/3 of healthcare costs provided for HF patients. The difficulty in treatment of patients with HF deterioration is associated with numerous comorbidities and coexisting complications (i.e. aggravation of ischaemic heart disease, lung diseases, infections, electrolyte disturbances, anaemia, renal failure as well as operations, in particular emergency ones). Our study is aimed to evaluation the complex pathophysiological background related to heart failure deterioration with respect to the effect of applied in-hospital treatment.

DETAILED DESCRIPTION:
PURPOSE:

Treatment of patients with heart failure (HF) is a great challenge for contemporary medicine. HF frequency in European population is assessed for 0.4 - 2%. This disease is characterized by high morbidity and mortality rate, poor quality of life and the necessity of frequent hospitalizations. Along with the medicine progress, in particular in the scope of acute coronary syndromes treatment, the number of HF patients is constantly growing. The essential problem connected with HF is its progress course and an increasing frequency of subsequent hospitalizations (approximately 30% of hospitalizations are the repeated ones). It is estimated that the costs of hospital stays constitute nearly 2/3 of healthcare costs provided for HF patients. In the United States approximately 50% of HF patients have been rehospitalized within 6 months from discharge and 70% of these hospitalizations were caused by HF deterioration.The prognosis in HF is closely connected with the progression of the disease defined in accordance with the NYHA (New York Heart Association) functional classification. The yearly mortality rate among each NYHA class is: class 1 - up to 10%, class 2 - 10-20%, class 3 - 20-40%, class 4 - mortality 40-60%. Over half of the patients with symptomatic HF die within 4 years of observation The high in-hospital mortality has been a great problem and results not only from the natural history of HF progression, but also from a number of coexisting complications (i.e. aggravation of ischaemic heart disease, lung diseases, infections, electrolyte disturbances, anaemia, renal failure as well as operations, in particular emergency ones). The optimal schemes of identifying the individual risk are of fundamental importance to guide the safe therapy. Undoubtedly hemodynamic status and its change during hospitalization is one of the main predictive factors of treatment response and occurrences of adverse effects of therapy, i.e. renal function worsening. However, there are no clear guidelines on how to perform safe and effective non-invasive hemodynamic monitoring.

AIMS:

The evaluation of complex pathophysiological features related to heart failure deterioration, including the parameters characterizing i.e. cardiovascular hemodynamics, hydration status, renal failure, iron metabolism and gas exchange, with respect to the effect of applied in-hospital treatment The evaluation of clinical value of the parameters characterizing i.e. cardiovascular hemodynamics, hydration status, renal failure, iron metabolism and gas exchange in prognosis of patients with heart failure deterioration

METHODS:

All the recruited patients will undergo the following assessment:

Clinical examination Laboratory tests, ncluding i.e. white blood cells count, red blood cells count, hemoglobin, hematocrit, mean cell volume (MCV), red cell distribution width (RDW); sodium, potassium, creatinine, estimated glomerular filtration rat (eGFR), urea, cystatin C; fasting glucose; bilirubin; total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglycerides, N-terminal of the prohormone brain natriuretic peptide (NT-proBNP); hs-TnT (high sensitive troponin T), iron; ferritin; unsaturated iron binding capacity (UIBC), total iron binding capacity (TIBC), transferrin saturation, soluble transferrin receptor; pH, carbon dioxide partial pressure (pCO2), oxygen partial pressure (pO2), arterial oxygen saturation (SaO2), bicarbonate content (HCO3-), base excess (BE), lactates; thyroid-stimulating hormone (TSH), testosterone, dehydroepiandrosterone sulfate (DHEAS), estradiol Electrocardiogram Echocardiography Chest X-ray Holter-ekg monitoring ambulatory blood pressure monitoring impedance cardiography (including assessment of: resting heart rate (HR), systolic and diastolic blood pressure (SBP and DBP), thoracic fluid content (TFC), cardiac index (CI), stroke index (SI), systemic vascular resistance index (SVRI) bioimpedance (including assessment total body water (TBW), intracellular and extracellular water (ICW, ECW)) applanation tonometry (including assessment of augmentation index (AI) and central pulse pressure (CPP))

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex
* urgent hospitalization caused by deterioration of HF.

Exclusion Criteria:

* unstable coronary artery disease including myocardial infarct within the last 40 days prior to recruitment
* stroke within 40 days prior to recruitment
* cardiac surgery within 90 days prior to recruitment
* pulmonary embolism
* severe pulmonary diseases (chronic obstructive pulmonary diseases - stage C/D, uncontrolled asthma, pulmonary hypertension)
* chronic kidney disease (stage 5 and requiring dialysis)
* severe inflammatory disease
* severe mental and physical disorders
* patients' refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure admitted to the Department of Internal Diseases and Cardiology urgently because of symptomatic heart failure deterioration
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-12; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
in-hospital death | 8 days
  time frame - assumed mean time of hospitalization
combined primary endpoint (in-hospital death and/or myocardial infract and/or stroke and/or serious arrhythmia and/or worsening renal function) | 8 days
  time frame - assumed mean time of hospitalization

SECONDARY OUTCOMES:
myocardial infract | 8 days
  time frame - assumed mean time of hospitalization
stroke (clinical symptoms and confirmed in CT) | 8 days
  time frame - assumed mean time of hospitalization
serious arrhythmia (new onset sustained ventricular tachycardia/fibrillation, supraventricular tachycardia, atrial fibrillation/flutter, sustained bradycardia <40/min) | 8 days
  time frame - assumed mean time of hospitalization
worsening renal function (increase in creatinine 0,3mg/dl according to the definition of AKDI) | 8 days
  time frame - assumed mean time of hospitalization

OTHER OUTCOMES:
significant electrolyte disturbances (K <3,0mmol/l; Na < 120mmol/l and or change in Na 10 mmol/l) | 8 days
  time frame - assumed mean time of hospitalization
symptomatic hypotension (SBP <90 mmHg or change in40 mmHg) | 8 days
  time frame - assumed mean time of hospitalization
hospitalization time (days) | 8 days
  time frame - assumed mean time of hospitalization
change in NYHA class | 8 days
  time frame - assumed mean time of hospitalization
"diuretic effectiveness ratio" - change in body mass change [%]/diuretics use [mg] | 8 days
  time frame - assumed mean time of hospitalization
change in HR | 8 days
  time frame - assumed mean time of hospitalization
change in SBP | 8 days
  time frame - assumed mean time of hospitalization
change in DBP | 8 days
  time frame - assumed mean time of hospitalization
change in SI | 8 days
  time frame - assumed mean time of hospitalization
change in CI | 8 days
  time frame - assumed mean time of hospitalization
change in TFC | 8 days
  time frame - assumed mean time of hospitalization
change in SVRI | 8 days
  time frame - assumed mean time of hospitalization
change in body mass | 8 days
  time frame - assumed mean time of hospitalization
change in TBW | 8 days
  time frame - assumed mean time of hospitalization
change in ECW | 8 days
  time frame - assumed mean time of hospitalization
change in ICW | 8 days
  time frame - assumed mean time of hospitalization
change in bilirubin | 8 days
  time frame - assumed mean time of hospitalization
change in eGFR | 8 days
  time frame - assumed mean time of hospitalization
change in urea | 8 days
  time frame - assumed mean time of hospitalization
change in hemoglobin | 8 days
  time frame - assumed mean time of hospitalization
change in hematocrit | 8 days
  time frame - assumed mean time of hospitalization
change in NTproBNP | 8 days
  time frame - assumed mean time of hospitalization
change in pH | 8 days
  time frame - assumed mean time of hospitalization
change in lactates | 8 days
  time frame - assumed mean time of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Krzesinski, MD, PhD, Principal Investigator — Military Institute of Medicine
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian Voivodeship, Poland